CLINICAL TRIAL: NCT01779661
Title: The Effect of Infant Aquatics for Neurodevelopment of Premature Infants
Brief Title: Infant Aquatics Neurodevelopment Premature Infants
Acronym: IA-NPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-12-9524-OB-CTIL
Record Dates: First submitted 2013-01-27; First posted 2013-01-30 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Cerebral Palsy; Preterm Birth; Development
Keywords: Neurodevelopment, Infant-Aquatics, Prematurity
MeSH Terms: conditions — Cerebral Palsy; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infant Aquatics (Active Comparator)
  Interventions: Other: Infant Aquatics
- Infant Massage (Active Comparator): Infant Massage
  Interventions: Other: Infant Massage

INTERVENTIONS:
Other: Infant Aquatics — Infant Aquatics in this study is composed of a set of pre-structured movements and techniques of relaxation, through harmonic integration of various approaches, each having a role in a specific time-window or in the infant's developmental sequence along study interventional timeline
  Arms: Infant Aquatics
Other: Infant Massage — Infant Massage
  Arms: Infant Massage

SUMMARY:
The objective of this research is to examine the effect of Infant Aquatics on the development of and neurodevelopment of preterm and near-term infants, using the GM as prognostic estimation of future development.

Preterm infants, a continuously growing population, are at high risk for neurodevelopment impairments ranging from minor neurological dysfunction (MND) to cerebral palsy (CP), mainly due to developmental brain injury. Infant Aquatics have been found to benefit and promote infant development. The support and sensory stimulation of the water may improve the development the sensory, motor, as well as, autonomic system of preterm infants.

The study will compare intervention by Infant Aquatics to infant massage. The intervention in both methods will start at 36 weeks gestational age for 3 months and will consist of sessions with a therapist every 2 weeks. Development will be assessed and compared at 3, 8 and 18 months using Infant Motor Pattern method, Griffith developmental scales and Vineland adaptive behavior scales.

ELIGIBILITY:
Inclusion Criteria:

Major inclusion criteria: Infants who are hemodynamic stable, no seizures or apnea attacks, IVH/PVH grade < 3, without diagnoses of chromosomal abnormalities, infants whose parents want to cooperate, will be included. These criteria follow our aim to include vulnerable groups of infants for which research results may dramatically promote development.

Exclusion Criteria:

infants whose parents are not able to understand research goals and refuse to cooperate, infants with seizures or apnea attacks, IVH/PVH grade >or =3, with diagnoses of chromosomal abnormalities.

Ages: 1 Week to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Developmental assessment - a composite of several measures | 3 month
  Developmental assessment at term and three month
  1. General Movements Neuromotor scale
  2. Neurological examination

SECONDARY OUTCOMES:
Developmental assessment - a composite of several measures | 18 month
  Developmental assessment at 18 month
  1. IMP neuromotor developmental scale
  2. Griffith mental development scale
  3. Vineland adaptive behavior scale

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Seba Medical Center, Ramat Gan, Israel